CLINICAL TRIAL: NCT00506571
Title: Phase II Study of S-1 Combined With Irinotecan and Oxaliplatin in Patients With Previously Untreated Metastatic Colorectal Cancer
Brief Title: Phase II Study of Irinotecan,Oxaliplatin Plus TS-1 in Untreated Metastatic Colorectal Cancer
Acronym: TIROX2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-07-261
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2007-04

CONDITIONS: Colorecal Neoplasms; Secondary
Keywords: colorectal neoplasms; secondary; Combination chemotherapy; S-1; irinotecan; oxaliplatin
MeSH Terms: conditions — Neoplasm Metastasis; Colorectal Neoplasms | interventions — S 1 (combination); Irinotecan; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: S-1, irinotecan, oxaliplatin

SUMMARY:
Patients will be treated with irinotecan (150 mg/m2) followed by oxaliplatin (85 mg/m2) on day 1 and S-1 (80 mg/m2/day) from day 1 to 14 every 3 weeks. Patients will receive up to a planned treatment of maximum 12 cycles of chemotherapy. Response assessment will be performed every 2 cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unresectable or metastatic colorectal cancer, not amenable to surgery or radiation treatment for curative intent
* At least one unidimensional measurable lesion
* ECOG performance status 0-2.
* No prior chemotherapy in metastatic settings, but adjuvant or neo-adjuvant treatment for non-metastatic (M0) disease is allowed if completed at least 6 months prior to initiation of study treatment
* Adequate major organ functions
* Give written informed consent

Exclusion Criteria:

* Prior systemic chemotherapy for metastatic disease
* Prior treatment with oxaliplatin or irinotecan
* Prior radiotherapy is permitted if it was not administered to target lesions selected for this study and provided it has been completed at least 4 weeks before registration
* Prior surgical treatment of stage IV disease is permitted
* CNS metastases
* Prior history of peripheral neuropathy ≥ NCI CTC grade 1
* Uncontrolled or severe cardiovascular disease
* Serious concurrent infection or nonmalignant illness
* Other malignancy within the past 3 years except cured non-melanomatous skin cancer or carcinoma in situ of the cervix
* Organ allografts requiring immunosuppressive therapy
* Psychiatric disorder or uncontrolled seizure that would preclude compliance
* Pregnant, nursing women or patients with reproductive potential without contraception
* Patients receiving a concomitant treatment with drugs interacting with S-1 such as flucytosine, phenytoin, or warfarin et al.
* Prior unanticipated severe reaction to fluoropyrimidine therapy, or known dihydropyrimidine dehydrogenase (DPD) deficiency
* Known hypersensitivity to platinum compounds or any of the components of the study medications
* Major surgery within 3 weeks prior to study treatment starts, or lack of complete recovery from the effects of major surgery
* Received any investigational drug or agent/procedure, i.e. participation in another trial within 4 weeks before beginning treatment with study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2007-07; Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Maximal overall response rate | During chemotherapy

SECONDARY OUTCOMES:
Progression-free survival, Overall survival, Toxicity assessment, & Pharmacokinetic characteristics and association with genetic polymorphism

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Hae Jung, M.D.Ph.D., Principal Investigator — not affiliated
Locations (1):
- National Cancer Center Korea, Goyang-si, Gyeonggi-do, South Korea